CLINICAL TRIAL: NCT03216187
Title: Swiss Multi-centre, Randomized, Placebo Controlled Trial of Pregabalin for Prevention of Persistent Pain in High Risk Patients Undergoing Breast Cancer Surgery
Acronym: PREVENT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient funding and recruitment
Sponsor: Benno Rehberg-Klug (Other)
Collaborators: University Hospital, Geneva (Other); Centre Hospitalier Universitaire Vaudois (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, médecin adjoint agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PREVENT
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Persistent Postoperative Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: study drugs (including identical placebos) and randomisation lists are prepared by the hospital pharmacy and are kept secret from the investigators until the end of the study and the "freezing" of the electronic data base (an interim analysis will be performed when data for the primary outcome are available for 60 patients per arm. Stopping rules are a difference in the incidence of the primary outcome of less than 8.2% (futility) or more than 19.9% (superiority)).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin 150 mg twice daily, starting from the evening before surgery, continuing with two times 150mg per day for 12 days, and ending with one 150mg capsule every evening for the final 3 days.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Identical placebo capsules twice daily, starting from the evening before surgery, continuing with two capsules per day for 12 days, and ending with one capsule every evening for the final 3 days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Pregabalin — pregabalin 150 mg capsules
  Other Names: Pregabalin 150mg capsules
  Arms: Pregabalin
Drug: Placebos — capsules identical to pregabalin but without active drug
  Other Names: placebo capsules
  Arms: Placebo

SUMMARY:
This study will test the benefits and risks of using pregabalin perioperatively to prevent persistent postoperative pain in patients at high risk (>30%) of developing such pain after breast cancer surgery.

DETAILED DESCRIPTION:
BACKGROUND Persistent postsurgical pain occurs in more than 30% of patients undergoing breast cancer surgery. Evidence that gabapentinoids such as pregabalin may reduce the incidence of persistent postsurgical pain is ambiguous, potentially because in previous trials prophylactic treatment was administered to every patient undergoing surgery. The patients at low risk of long term pain, were exposed to side effects without much benefit to expect.

AIM Validating or refuting the utility of pregabalin to prevent long term post-operative pain in patients at high risk of persistent pain after breast cancer surgery.

METHODS Randomized, double-blind, placebo-controlled trial of pregabalin (2*150mg from the day before breast cancer surgery until 2 weeks after surgery) in patients at high risk of persistent pain (>30%). High-risk patients are identified by a risk score derived from a previous observational study. The main outcome is the incidence of clinically important pain (necessitating analgesic treatment, or having an intensity of >3 at rest or >5 on movement) at 3 months after surgery. Secondary outcomes are: incidence of neuropathic pain, pain interference, and incidences at 6 and 12 months of follow-up. In addition, side effects of pregabalin and the retention rate during the treatment period will be monitored, as well as patient expectancies.

RELEVANCE This is the first study for prevention of persistent postoperative pain which targets only high-risk patients, thus lowering a false negative outcome and averting the risk of side effects for patients at low risk.

The study is powered to show a reduction of the incidence of clinically important pain at 3 months of 20%. In the case the study shows that this can be achieved and pregabalin is well tolerated, the preventive use of pregabalin for breast cancer surgery would be justified at least in high-risk patients. On the other hand, a negative result would indicate the futility of pregabalin prevention, which is already in routine use in many hospitals.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for breast surgery for cancer, either breast-conserving (tumorectomy/ quadrantectomy) or mastectomy, with or without immediate reconstruction, and with or without axillary dissection.
* patients of 18 years or more scheduled for above mentioned type of surgery
* ability to speak and read French, English or German
* high (>30%) risk of clinically important persistent pain: identified with 2 or more points of a risk score including the items: pre-existing pain at surgical site (2 points), history of depression (1 point), age < 50 years (1 point), and high expected acute pain (>6/10, 1 point).
* Informed Consent as documented by signature.

Exclusion Criteria:

* Inability to understand the consent form and to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Pregnancy or lactation - Renal insufficiency (creatinine clearance < 60 ml/min)
* Allergy to pregabalin or the ingredients of the capsules
* Long-term preoperative therapy with gabapentinoids or high-dose opioids (more than 60 mg of morphine equivalents)
* Symptomatic cardiac insufficiency (peripheral oedema, NYHA class III - marked limitation of physical activity)
* Suicidal ideation, identified by the question: "have you been bothered by thoughts that you would be better off dead, or of killing yourself?"
* Planned fertility preservation immediately after surgery before a planned chemotherapy
* Known or suspected non-compliance, or substance-use disorder with impact on medication adherence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
incidence of "clinically important pain" at 3 months after surgery | 3 months
  "Clinically important pain" is defined by: taking analgesics for pain at the surgical site OR average resting pain at the surgical site >3/10 OR average movement-induced pain at the surgical site >5/10.

SECONDARY OUTCOMES:
Pregabalin-related side effects | 10 days
  blurred vision or diplopia, somnolence or sleepiness, abnormal thinking, confusional state, disturbed attention, and falls, as well as the effects noted in the "generic assessment of side effects" GASE questionnaire
retention rates of pregabalin treatment | 30 days
acute pain intensity and patient-reported pain outcome at 24h | 24 hours
  PAIN-OUT questionnaire
pain intensity at rest and movement, pain interference | 3, 6, and 12 months
  Brief Pain Inventory, BPI
neuropathic pain | 3, 6, and 12 months
  incidence of neuropathic pain defined as a DN4-self-evaluation score ≥4
patient-reported relevance of pain | 3, 6, and 12 months
  response to the question: "do you consider your pain as significant?"
Patient-reported acceptance of the preventive treatment | 3 months
  response to the question "In retrospect, do you consider the preventive treatment worthwhile, given your pain outcome and your experience of taking the medication?")
Expectations about treatment benefits before treatment and after | 10 days
  responses to the questions: "How much pain do you expect 3 months from now?"" "How efficient do you think the study treatment is against the long-term pain (i.e. what is the success rate in %)?" "How well do you think it will work for you? (i.e. reduction in pain score 0-10)". Beliefs about treatment attribution after 10 days of treatment (question: "Do you think that you received the real drug or the placebo?")

CONTACTS AND LOCATIONS:
Overall Officials: Benno Rehberg-Klug, MD, Study Director — HUG; Marc Suter, MD, Study Director — CHUV; Ulrike Stamer, MD, Study Director — Inselspital
Locations (6):
- Switzerland (6):
  - Inselspital, Bern
  - Brustzentrum Bern, Bern
  - Hôpitaux Universitaires de Genève HUG, Geneva
  - Clinique des Grangettes, Geneva
  - Clinique de Genolier, Genolier
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne

IPD SHARING:
Plan to Share IPD: Undecided